CLINICAL TRIAL: NCT06527261
Title: Electronic Capturing of Activities During REhabilitation for Upper Limb After Stroke
Acronym: eCARE4Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Other Study IDs: HREC/107078/Austin-2024
Record Dates: First submitted 2024-07-11; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Usual care; Upper extremity; Dose; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Sessions: Observed sessions for patients who are in the acute inpatient setting. Each session will include a patient and a clinician
  Interventions: Other: Real-time electronic data input into REDCap
- Subacute Sessions: Observed sessions for patients who are in the subacute inpatient setting. Each session will include a patient and a clinician
  Interventions: Other: Real-time electronic data input into REDCap

INTERVENTIONS:
Other: Real-time electronic data input into REDCap — During usual care sessions, clinicians will real-time capture information about the intervention session into REDCap. This information is related to the multi-dimensional dose articulation framework e.g., content of the session and difficulty of the task, session length, episode length, and number of repetitions.
  The usual care motor upper limb intervention the patient receives is determined by the clinician providing the care. The therapy may include but is not limited to strength training, task specific retraining, constraint induced movement therapy, mirror box, and electrical stimulation.

SUMMARY:
This is a prospective cohort study to determine the feasibility of accurate, complete, and timely real-time electronic capturing of upper limb motor intervention sessions during usual care. In clinical trials accurate reporting of usual care for people with stroke is scarce, thus understanding the control group compared to the experimental group is poor. The unit of measure in this study is therapy sessions, where a clinician is providing usual care to a patient.

The observed sessions will occur in two Austin Health settings: Acute at Austin Hospital; subacute, across Royal Talbot Rehabilitation Centre or the Heidelberg Repatriation Hospital. For each session, patient characteristics, dose and content of upper limb interventions will be electronically captured in REDCap. Additionally, the sessions will be video recorded to allow a second rater to assess feasibility. The secondary aim is to determine if there is an association between the dose and content of upper limb intervention sessions and the contextual factors of stroke patients. Two participant groups will be recruited: Stroke patients and Clinicians (Occupational Therapists and Allied Health Assistants).

DETAILED DESCRIPTION:
This is a prospective observational cohort study to determine the feasibility of accurate, complete, and timely real-time electronic capturing of upper limb motor intervention sessions during usual care.

In clinical trials accurate reporting of usual care for people with stroke is scarce, thus understanding the control group compared to the experimental group is poor.

The unit of measure is the therapy sessions, where a clinician is providing usual care to a patient. The observed sessions will occur across two Austin Health settings. Setting A: Acute at Austin Hospital, and Setting B: Subacute at Royal Talbot Rehabilitation Centre or the Heidelberg Repatriation Hospital.

For each session, patient characteristics, the multiple dimensions of dose, and the content of usual care motor upper limb interventions will be electronically captured in REDCap. The observed sessions will be video recorded and a second rater will review the session for dose data accuracy. Secondary to determining feasibility, the dose and content data from observed sessions will be analysed to investigate the association of context factors such as setting and upper limb impairment severity.

As such, this study aims to answer the following research questions:

* Is it feasible for clinicians to electronically capture accurate, complete, and timely upper limb motor intervention session dose during usual care of stroke patients?
* Is there an association between dose and content of upper limb intervention sessions and the contextual factors of stroke patients?

ELIGIBILITY:
Group 1: Stroke patients

Inclusion Criteria:

* Adults (≥18 years) with a new, first or consecutive stroke, confirmed on CT or MRI.
* Motor upper limb impairment defined by a Shoulder Abduction and Finger Extension (SAFE) score of 0 through 9.
* Able to consent for themselves.
* Likely to receive at least one upper limb intervention session as determined by the treating clinical team.

Exclusion Criteria:

* Existing co-morbidities that limit upper limb function and usual care treatment provided as determined by the treating clinical team e.g., neural or orthopeadic
* Receiving palliative care or have a limited life expectancy
* Deemed unable or unnecessary to participate in upper limb intervention by the treating clinical team
* Treating Occupational Therapist and local allied health assistant declined to participate in the research preventing recording of usual care data
* Unable to follow basic instructions in English

Group 2: Clinicians

Inclusion criteria

* Occupational therapist or allied health assistant working with the stroke population in an acute or subacute settings within Austin Health.
* At least four months of clinical experience

Exclusion criteria:

• Clinicians expected to move into another clinical area within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Stroke patients These participants will be selected from inpatients within the tertiary health service of Austin Health in Melbourne, Victoria, Australia. They may be located at the acute setting: Austin hospital, Or subacute setting: Heidelberg repatriation hospital or Royal Talbot rehabilitation Centre.
  Group 2: Clinicians Clinicians will be invited to participate if they are an Occupational Therapist or allied health assistant working at Austin health with the stroke patient population.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of real-time electronic data input of usual care session dose | Each feasibility session will take up to one hour.
  A single binary composite primary outcome, where feasibility is defined by 90% of sessions achieving ALL of:
  1. Binary outcome of Accuracy: ≤10% difference in dose between electronic data and second-rater data from a video recording of the session as defined by the decision algorithm.
  2. Binary outcome of Completeness: ≥90% of the electronic data completed by clinicians as defined by the decision algorithm.
  3. Binary outcome of Timeliness: ≤10% of session time is spent completing the electronic record or rated non-burdensome by the clinician as defined by the decision algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hayward, Principal Investigator — University of Melbourne
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No